CLINICAL TRIAL: NCT02489513
Title: A Phase 1, Open-label Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-AG-120 Following Single Oral Dose Administration in Healthy Male Subjects
Brief Title: Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-AG-120
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AG120-C-003
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group assignment (Other): [14C]-AG-120
  Interventions: Drug: [14C]-AG-120

INTERVENTIONS:
Drug: [14C]-AG-120 — Labeled investigational drug

SUMMARY:
The study is designed to characterize the absorption, metabolism, and excretion of AG-120 using radiolabeled drug in healthy adult male subjects to support its further development and registration.

DETAILED DESCRIPTION:
This will be a single-center, open-label, study in healthy adult males. Each subject will participate in a screening phase, a baseline phase, a treatment phase, and a follow up period. Subjects who have met all inclusion criteria and none of the exclusion criteria at screening will return to the clinical site on Day -1 for baseline assessments. Following a 10 hour overnight fast, subjects will receive a single 500mg dose of AG-120 suspension containing a microtracer of [14C] AG-120 (~ 200 μCi) under fasted conditions. The study drug will be administered as an oral suspension with approximately 240 mL of room temperature, non-carbonated water.

Blood, urine, and fecal samples (and vomitus, if applicable) will be collected throughout the study for pharmacokinetic (PK), mass balance, and/or clinical laboratory assessments. Safety will be monitored throughout the study. Subjects will be discharged from the clinical site from Day 22 to Day 29, depending on the recovery of eliminated radioactivity.

Urine and fecal samples will be collected each day until Day 29 (or the point of discharge if earlier) for measurement of total [14C] radioactivity. Blood samples for radioanalysis and PK assessment, inclusive of metabolite profiling/characterization, will be collected at pre-dose and at specified intervals through Day 29. Total [14C]-radioactivity in whole blood, plasma, urine, and feces (and vomitus, if applicable ) will be determined.

Up to 8 subjects will enroll in the study. One to two additional subjects who have been confirmed as having poor metabolizer (PM) CYP2D6 genotype may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy adult male of any race and aged 18 to 55 years, inclusive, at the time of signing the Informed Consent Form (ICF)
2. Understands and voluntarily signs an ICF before any study-related assessments/procedures are conducted
3. Is willing and able to adhere to the study visit schedule and other protocol requirements
4. Is willing to provide a blood sample for genotyping of CYP2D6 status at Screening
5. Is either sterile or agrees to use contraception from Check-in until 90 days following dose administration. The approved methods of contraception include: male condom with spermicide (foam, gel, film, cream, or suppository); sterile sexual partner (eg, tubal occlusion, hysterectomy, or bilateral salpingectomy); or by female sexual partner, established use of hormonal contraceptives, use of an intrauterine device with copper or intrauterine system with progestogen, barrier contraceptive (condom, diaphragm, or cervical/vault caps) used with spermicide, or true abstinence; periodic abstinence (eg, calendar, ovulation, symptothermal post-ovulation methods) is not an acceptable method of contraception.
6. Must have a body mass index between 18 and 33 kg/m2, inclusive, at Screening
7. Must be healthy as determined by the Investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead ECG at Screening

   * Must be afebrile (febrile is defined as ≥38.5°C or 101.3°F)
   * Supine systolic blood pressure (BP) must be in the range of 90 to 140 mmHg, supine diastolic BP must be in the range of 50 to 90 mmHg, and pulse rate must be in the range of 40 to 110 beats per minute, as confirmed by repeat assessment if the initial vitals are out of range
   * Normal or clinically acceptable 12-lead ECG, with a QT interval corrected using Fridericia's formula (QTcF) value ≤430 msec
   * Calcium, magnesium, and potassium levels within normal ranges

Exclusion Criteria:

1. History of any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
2. Any condition, including the presence of clinically significant laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study
3. Any condition that confounds the ability to interpret data
4. Exposure to an investigational drug (new chemical entity) within 30 days preceding dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer)
5. Participation in more than 1 other radiolabeled investigational drug study within 12 months prior to Check-in (Day -1)
6. Significant radiation exposure (eg, serial X-ray or computed tomography scans, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in (Day -1)
7. Prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc.) within 30 days of dose administration
8. Nonprescription systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of dose administration
9. Received a live vaccination within 90 days of dose administration
10. Surgical or medical conditions possibly affecting absorption, distribution, metabolism, or excretion, (eg, bariatric procedure, or plans to have elective or medical procedures performed during the conduct of the trial). Prior appendectomy is acceptable, but prior cholecystectomy would result in exclusion from the study
11. Blood or plasma donation within 8 weeks before dose administration to a blood bank or blood donation center
12. History of drug abuse within 2 years before dose administration, or positive drug screening test reflecting consumption of illicit drugs
13. History of alcohol abuse within 2 years before dose administration, or positive alcohol screen at Check-in
14. Use of any tobacco- or nicotine-containing products (including but not limited to cigarettes, e-cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to Screening, or positive cotinine screen
15. Known to be a carrier of hepatitis B surface antigen or hepatitis C virus antibody, or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening
16. Employed by the clinical site, or is related to an employee of the clinical site
17. History of less than 1 bowel movement per day

Standard dietary, fluid intake, and exercise restrictions are required as part of the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Total [14C] Whole blood and plasma | up to 29 days
  Total [14C]-radioactivity in whole blood and plasmafollowing oral administration of a single 500-mg (approximately 200 μCi) radiolabeled dose of AG-120 in male subjects
Pharmacokinetics of single dose of AG-120 (Cmax) | up to 29 days
  time of maximum observed drug concentration
Pharmacokinetics of single dose of AG-120 (AUC) | up to 29 days
  Area under the curve
Pharmacokinetics of single dose of AG-120 (t1/2) | up to 29 days
  Estimate of the terminal elimination half-life
Pharmacokinetics - Total [14C] urine and feces | up to 29 days
  Total [14C]-radioactivity in urine, and feces (and vomitus, if applicable).

SECONDARY OUTCOMES:
AG120 Metabolite identification | up to 29 days
  Blood, urine, and fecal sample analysis to identify metabolites of AG-120

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Agresta, MD, MPH, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- Research Site, Madison, Wisconsin, United States